CLINICAL TRIAL: NCT00489580
Title: A Pilot Study Investigating the Feasibility of Using a Functional Tone Management (F.T.M.) Arm Training Program With the SaeboFlex Dynamic Hand Orthosis on an Inpatient Population
Brief Title: A Pilot Study Investigating the Feasibility of the Saebo Arm Training Program on an Inpatient Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: Saebo, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-519-05
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Stroke; Hemiplegia
Keywords: stroke; weakness; motor recovery
MeSH Terms: conditions — Stroke; Hemiplegia; Asthenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SaeboFlex Dynamic Hand Orthosis
Procedure: Saebo F.T.M. Arm Training Program

SUMMARY:
Study Objectives:

1. To document the safe and effective application of the F.T.M. Arm Training Program using the SaeboFlex to an inpatient post stroke rehabilitation population.
2. To compare functional improvements in hand and UE use achieved with the F.T.M. program as compared to generally applied therapeutic treatment approaches.
3. To develop recommendations for an inpatient retraining protocol that could then be evaluated in a multi-center trial.
4. To document the retention of UE and hand improvements after SaeboFlex training is discontinued as well as the carry over of these gains into daily function after therapy has been discontinued.

DETAILED DESCRIPTION:
Therapeutic interventions for the recovery of hand function after a neurological injury have historically been very limited. A significant body of research now supports the use of an upper extremity retraining approach for functional recovery after neurological injury. Few therapeutic approaches offer any intervention specifically focused on grasp and release retraining. In an effort to address this deficit, the SaeboFlex dynamic hand orthosis was developed by occupational therapists. The F.T.M. Arm Training Program has been safely used by hundreds of occupational and physical therapists on over one thousand patients in outpatient neurological rehabilitation over the past two years. It is currently an accepted modality of treatment for the management of hand paresis in the acquired brain injury population. During that time, two factors, other than the severity of the initial injury, were identified as having a significant affect on the outcomes achieved in treatment. They are learned non-use and soft tissue shortening of the finger flexors. All treatment delivered to the subjects that partake in this study will be clinical care and the only research component of this study will be the assessment of outcomes. The purpose of this study is to explore the proper treatment dosage and treatment protocol for the application of the F.T.M. Program to the inpatient post stroke rehabilitation population. Additionally, information on functional outcome measures will be collected and compared to a matched control group that undergoes the standard therapeutic protocol.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Must be seen within three full working days of admission for screening
* Alert and Oriented to person and place with the ability to complete at a minimum a one step verbal command,
* Demonstrated active range of motion of 10 degrees shoulder flexion / abduction and 10 degrees of elbow flexion / extension
* 1/4 range of volitional finger flexion when the affected hand is passively positioned in a minimum of 15degrees of wrist extension with the MCP's at neutral and PIP's / DIP's in extension
* Patient must be independent with seated posture in a chair with a firm seat and back support but no arm rests
* Patient can maintain independent seated balance when unaffected upper extremity is fully outstretched in any direction
* Admitted to inpatient stroke rehabilitation at Kessler Institute

Exclusion Criteria:

* Inpatient physician unwilling to clear patient to participate
* Medically unsuitable for therapeutic intervention,
* Using the affected hand and arm, able to volitionally grasp and release a racquet ball x10 at maximal volitional shoulder flexion with wrist extension of 10 degrees or more.
* Flaccidity in the affected UE or hand
* Fixed joint deformities, contractures or joint hypermobility that prevents proper joint positioning in the orthosis.
* Hx of rheumatoid arthritis, carpal tunnel syndrome or other hand neuropathy
* Moderate to severe weeping or pitting edema
* No previous stroke prior to the one prompting admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-08; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Hand grip strength (measured using dynamometry) | At admission and at discharge

SECONDARY OUTCOMES:
Length of Stay (days) | The duration of the subject's inpatient hospital stay.
Stroke Impact Scale Score | At admission and at discharge
Action Research Arm Test Score | At admission and at discharge
Ashworth Assessment (Upper Extremity) Scores | At admission and at discharge
Fugl-Meyer Assessment (Upper Extremity) Scores | At admission and at discharge
Goniometric Range of Motion Evaluation, Passive and Active (Shoulder, Elbow, and Wrist) | At admission and at discharge
Assessment of Active Range of Motion (Fingers, as ¼ range, ½ range, ¾ range or full range) | At admission and at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Elie P Elovic, M.D., Principal Investigator — Kessler Medical Rehabilitation Research & Education Center
Locations (1):
- Kessler Institute for Rehabilitation, East Orange, New Jersey, United States